CLINICAL TRIAL: NCT02461576
Title: Clinical Evaluation of the Xpert® HIV-1 VL: A Method Comparison Study
Brief Title: Clinical Evaluation of the Xpert® HIV-1 VL
Status: Completed | Type: Observational
Sponsor: Cepheid (Industry)
Responsible Party: Sponsor
Other Study IDs: 177B
Record Dates: First submitted 2015-05-26; First posted 2015-06-03 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV-1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Leftover plasma specimens will be retained in a biobank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1 infected: this is a study comparing Xpert HIV-1 VL assay quantitation to an already FDA approved HIV-1 quantitative HIV-1 RNA assay in known HIV-1 infected individuals
  Interventions: Device: Xpert HIV-1 VL Assay

INTERVENTIONS:
Device: Xpert HIV-1 VL Assay — in vitro diagnostic test to quantify HIV-1 RNA

SUMMARY:
Compare the clinical performance of the Xpert® HIV-1 VL to another FDA approved HIV-1 RNA quantitative assay using frozen and fresh specimens from known HIV-1 positive individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositive adults using an FDA approved method
* At least 18 years of age or older
* Informed consent, if applicable

Exclusion Criteria:

* Subject is less than 18 years of age
* Previously enrolled in this study
* Samples not collected according to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females >18 yours who are known HIV-1 infected and may be on treatment or untreated with ARV therapy
Sampling Method: Non-Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Quantification of HIV-1 RNA in copies/mL in known HIV-1 positive subjects | 1 day (A single time point)
  This study is a comparative analysis of HIV-1 RNA quantitation between Xpert HIV-1 VL to another FDA approved test. A single time point (cross-sectional) from each of at least 300 subjects with HIV-1 RNA quantitation within the dynamic range of both assays will be used in regression models to assess performance of the Xpert HIV-1 VL in comparison to the other FDA approved test.